CLINICAL TRIAL: NCT04106401
Title: Alterations in Total Red Blood Cell Volume and Plasma Volume During a One-year Confinement in Antarctica: Effect of Hypoxia
Brief Title: Intravascular Volumes in Hypoxia During Antarctic Confinement
Acronym: ANTARCV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ecole Nationale des Sports de Montagne (Other)
Collaborators: Center for Physical Activity Research, University Hospital of Copenhagen, Denmark (Unknown); Laboratory Mobility, aging & exercise (MOVE) -EA 6314, Faculty of Sport Sciences, University of Poitiers, France (Unknown); Department for Biomedical Sciences for Health, University of Milan School of Medicine, Milan, Italy (Unknown); HP2 Laboratory, INSERM, Grenoble Alpes University, CHU Grenoble Alpes, Grenoble, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A03243-52
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Hypoxia; Confinement
Keywords: total red blood cell volume; plasma volume; total hemoglobin mass; total blood volume
MeSH Terms: conditions — Hypoxia | interventions — Blood Specimen Collection; Blood Pressure

STUDY DESIGN:
Intervention Model Description: one group wintering at sea level and one group wintering at high altitude
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypoxia & confinement (Experimental): Participants exposed to high-altitude hypoxia and confinement during a one-year stay at Concordia station, Antarctica (3200 m)
  Interventions: Other: carbon-monoxide rebreathing; Other: venous blood sampling; Other: physical activity monitoring; Other: apnea-hypopnea index and nocturnal oxygenation; Other: 24-hour blood pressure
- confinement (Active Comparator): Participants exposed to confinement during a one-year stay at Dumont d'Urville station, Antarctica (sea level)
  Interventions: Other: carbon-monoxide rebreathing; Other: venous blood sampling; Other: physical activity monitoring; Other: apnea-hypopnea index and nocturnal oxygenation; Other: 24-hour blood pressure

INTERVENTIONS:
Other: carbon-monoxide rebreathing — Inhaled carbon monoxide (CO) administrated as a bolus into a rebreathing circuit serves as a marker to tag circulating hemoglobin molecules and to calculate total hemoglobin mass (Hbmass). The change in blood CO concentration from pre- to postadministration (delta carboxyhemoglobin concentration) and the dose of administrated CO allows for Hbmass determination. The other blood compartments (total red blood cell volume, plasma volume and total blood volume) are derived from Hbmass, hematocrit and/or hemoglobin concentration.
Other: venous blood sampling — venous blood sampling at rest to evaluate blood viscosity, erythropoiesis and iron metabolism
Other: physical activity monitoring — recording of physical activity by actimetry
Other: apnea-hypopnea index and nocturnal oxygenation — recorded by ambulatory sleep recording device
Other: 24-hour blood pressure — recorded by ambulatory device

SUMMARY:
This study evaluates the effect of hypoxia on blood volumes during Antarctic winter-over confinement. Half of the participants will be evaluated during sea-level winter-over confinement, while the other half will be examined during high-altitude hypoxia winter-over confinement.

DETAILED DESCRIPTION:
INTRODUCTION: Short-term space flight induces an alteration of circulating blood volumes, termed "space flight anemia" and characterized by a decrease in total red blood cell volume (RCV) and plasma volume (PV). This haematological alteration is likely to persist during a long-term space mission and impact the astronauts' health, however this question remains unexplored. During a long-term space mission, the use of hypobaric hypoxia is considered for technical reasons, however the safety of hypoxia must first be verified because this environmental condition causes substantial physiological changes, in particular changes in blood volumes that may interact with the haematological effects of microgravity.

OBJECTIVE: using the Antarctic confinement model as a high-fidelity terrestrial analogue for long-duration space missions, the investigators hypothesize that 1) sea level confinement reduces blood volume by simultaneously decreasing RCV and PV, and 2) chronic hypoxia offsets the decrease in RCV and exacerbates the decrease in PV induced by confinement.

METHODS: blood volumes will be measured via the carbon-monoxide rebreathing method, repeatedly in two groups of participants, overwintering either at Dumont d'Urville (sea level) or Concordia (altitude 3200 m). The blood viscosity will also be measured, as well as the markers of erythropoiesis and iron metabolism.

PERSPECTIVE: Documenting if some degree of hypoxia during long-duration confinement may be beneficial or unfavorable in terms of blood volume regulation is potentially relevant information for the astronauts' health and safety during long-duration space missions.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a social security scheme
* Ability to communicate and read in English or in French
* Signed written informed consent form after visit with a MD

Exclusion Criteria:

* Pregnant, lactating or parturient women
* Cardiovascular, pulmonary or neuromuscular disease
* Vulnerable persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
total hemoglobin mass | 15 months
  Physiological parameter, corresponding to the total amount of circulating hemoglobin, expressed in grams, and determined with the 10-min carbon-monoxide rebreathing method and blood carboxyhemoglobin measurements (expressed in %).
total red blood cell volume | 15 months
  Physiological parameter, corresponding to the total volume of circulating red blood cells, expressed in liters, and derived from total hemoglobin mass, hematocrit (expressed in fraction) and hemoglobin concentration (expressed in gram per deciliter).
total blood volume | 15 months
  Physiological parameter, corresponding the the total volume of blood, expressed in liters, and derived from total red blood cell volume and hematocrit.
plasma volume | 15 months
  Physiological parameter, corresponding to the total volume of plasma, expressed in liters, and derived from total blood volume and total red blood cell volume.

SECONDARY OUTCOMES:
blood viscosity | 15 months
  Physiological parameter, corresponding to the dynamic viscosity of whole blood, expressed in centipoises, and determined by a cone/plate viscometer
serum erythropoietin | 15 months
  Physiological parameter, corresponding to the serum concentration of erythropoietin expressed in milli-International unit per ml, determined by a specific biological assay.
serum hepcidin | 15 months
  Physiological parameter, corresponding to the serum concentration of hepcidin, expressed in mmol per liter, determined by a specific biological assay.
serum erythroferrone | 15 months
  Physiological parameter, corresponding to the serum concentration of erythroferrone, expressed in ng per ml, determined by a specific biological assay.
serum transferrin saturation | 15 months
  Physiological parameter, corresponding to the serum transferrin saturation, expressed in %, derived from serum iron concentration (in µg/dl) and transferrin concentration (in mg/dl)
serum ferritin | 15 months
  Physiological parameter, corresponding to the serum concentration of ferritin, expressed in ng per ml, determined by a specific biological assay.
serum soluble transferrin receptor | 15 months
  Physiological parameter, corresponding to the serum concentration of soluble transferrin receptor, expressed in nmol per liter, determined by a specific biological assay.
Physical activity | 15 months
  Physiological parameter, corresponding to the level of daily energy expenditure, expressed in kilocalories per kg per day, determined by accelerometry.
Apnea-hypopnea index | 15 months
  Physiological parameter, corresponding to apnea-hypopnea events, expressed in events per hour, recorded by an ambulatory sleep recording device.
Nocturnal oxygenation | 15 months
  Physiological parameter, corresponding to pulse oxygen saturation, expressed in %, recorded by an ambulatory sleep recording device.
24-hour blood pressure | 15 months
  Physiological parameter, corresponding to the mean arterial blood pressure over 24 hours, expressed in mmHg, recorded by an ambulatory device

CONTACTS AND LOCATIONS:
Locations (1):
- Ecole nationale des sports de montagne, site de l'Ecole nationale de ski et d'alpinisme, Chamonix, Haute Savoie, France

IPD SHARING:
Plan to Share IPD: No